CLINICAL TRIAL: NCT05462210
Title: The Effect of Mobilization Protocol Assisted With Simulated Clinical Immersion Videos on Postoperative Pain, Fear of Movement, Mobility Level and Satisfaction in Patients Undergoing Lumbar Spine Surgery: A Randomized, Controlled, Single-Blind Study
Brief Title: The Effect of Mobilization Protocol Assisted With Simulated Clinical Immersion Videos on Patients Undergoing Lumbar Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Arş. Gör. Arzu TAT ÇATAL, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KAEK-312
Record Dates: First submitted 2022-06-30; First posted 2022-07-18 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Lumbar Spine Surgery; Lumbar Disc Herniation
Keywords: Mobilization; Nursing; Spinal Surgery; Pain; Fear of Movement; Patient Satisfaction; Simulation
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain; Kinesiophobia; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants and statistician are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The first mobilization of patients undergoing surgical treatment for lumbar disc herniation in the clinics where the study will be conducted is routinely performed within the first 24 hours after surgery. When the data collection process of the control group is completed, the data will be integrated with the mobilization protocol assisted with simulated clinical immersion videos created for the research.
- Intervention group (Experimental): Mobilization Protocol Assisted with Simulated Clinical Immersion Videos Simulated clinical immersion videos created for the mobilization protocol for patients in the intervention group will be sent to their smartphones once they are admitted to the clinic. The videos prepared within the scope of the mobilization protocol will be watched by patients in company with the researcher the day before the operation, their questions will be answered, and the correct mobilization techniques will be shown practically. It is expected that patients watch the videos at least four times, as twice with the researcher and twice by themselves.
  Interventions: Other: Mobilization Protocol Assisted with Simulated Clinical Immersion Videos

INTERVENTIONS:
Other: Mobilization Protocol Assisted with Simulated Clinical Immersion Videos — Mobilization Protocol Assisted with Simulated Clinical Immersion Videos Simulated clinical immersion videos created for the mobilization protocol for patients in the intervention group will be sent to their smartphones once they are admitted to the clinic. The videos prepared within the scope of the mobilization protocol will be watched by patients in company with the researcher the day before the operation, their questions will be answered, and the correct mobilization techniques will be shown practically. It is expected that patients watch the videos at least four times, as twice with the researcher and twice by themselves.
  Arms: Intervention group

SUMMARY:
This study focused on examining the effect of mobilization protocol assisted with simulated clinical immersion videos on postoperative pain, fear of movement, mobility level and satisfaction in patients undergoing lumbar spine surgery.

DETAILED DESCRIPTION:
Background: The medical condition that creates the need for lumbar spine surgery causes pain and movement restriction in patients. Ensuring safe mobilization in patients with lumbar spine surgery is important for pain management and prevention of complications.

Aim: In this study, it was aimed to examine the effect of mobilization protocol assisted with simulated clinical immersion videos on postoperative pain, fear of movement, movement level and satisfaction.

Study Design: The study was designed as interventional, pre-test, post-test, parallel group, single-blind, randomized, controlled and experimental. In the study, patients in the control group will be applied routine protocols, and patients in the intervention group will be trained on the day before surgery using the mobilization protocol assisted with simulated clinical immersion videos. In this study, the patients will be distributed to the groups by the "block randomization method".

Methods: In this study, pain, fear of movement, movement level and satisfaction will be recorded at the first postoperative mobilization and discharge.

ELIGIBILITY:
Inclusion Criteria:

* According to the ICD-10 Codes: Those with S33.0-Traumatic rupture of lumbar intervertebral disc, G55-Nerve root and plexus compressions, M54.4-Lumbago with sciatica, underwent lumbar disc herniation surgery (microdiscectomy) due to diagnosed with M54.5-Low back pain,
* Aged 18 and over,
* With no hearing, vision, comprehension and speech impairments,
* Volunteering to participate in the research,
* Using a smartphone will be included in the study.

Exclusion Criteria:

* Those under the age of 18,
* Underwent revision lumbar spine surgery,
* With mental or physical disabilities to receive the mobilization training that will be provided before the operation will not be included in the sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Back and leg pain | Changes in hospitalization, first mobilization after surgery and the day of discharge. 1. Day of hospitalization (24 hours) 2. The first 24 hours after surgery 3. The day of discharge (24 hours)
  The Visual Analog Scale (VAS) is a straight horizontal line of 100 mm. One end describes no paint at all while the other describes an excessive amount of pain. VAS score is calculated by measuring in millimeters from the left end of the line to the point marked by the patient. VAS will be used to assess low back pain (VAS-BP) and right and left leg pain (VAS-LP) separately (Nayak, Coats, Abdullah, Stein, & Malhotra, 2015).
Fear of Movement | Changes in hospitalization, first mobilization after surgery and the day of discharge. 1. Day of hospitalization (24 hours) 2. The first 24 hours after surgery 3. The day of discharge (24 hours)
  Tampa Scale for Kinesiophobia (TKS): The TKS is used to assess the subjective degree of kinesiophobia or fear of movement, and consists of 17 items. The 4-point Likert-type scale ranges from 1 to 4 (1=Strongly disagree, 4=Completely agree). The overall score is calculated after reverse scoring the items 4, 8, 12 and 16. The overall scale score ranges between 17 and 68, and higher scores indicate higher level of kinesiophobia (Yılmaz et al., 2011).
Mobility Level | Changes in hospitalization, first mobilization after surgery and the day of discharge. 1. Day of hospitalization (24 hours) 2. The first 24 hours after surgery 3. The day of discharge (24 hours)
  Patient Mobility Scale: The level of pain and difficulty that patients experience doing four activities (turning from side to side in bed, sitting on the edge of the bed, sitting up at the side of the bed, walking in hospital room) during the postoperative period are assessed using a 15-cm visual analogue, throughout which verbal expressions are included. The lowest and highest possible scores obtained from each item ranges between 0 and 15, and the overall scale score ranges between 0 and 120. Higher scores indicate higher level of pain and difficulty (Ayoğlu, 2011).

SECONDARY OUTCOMES:
Patient Satisfaction | The day of discharge (24 hours)
  Patients' satisfaction with the care they receive will be assessed using a Visual Analog Scale. The Visual Analog Scale (VAS) is a straight horizontal line of 100 mm. One end describes not satisfied at all, while the other describes high level of satisfaction. VAS score is calculated by measuring in millimeters from the left end of the line to the point marked by the patient. Higher scores indicate higher level of satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)